CLINICAL TRIAL: NCT02215590
Title: Re-Step: a Computerized Dynamic Balance Treatment for Rehabilitation of Unassisted Gait in ABI Victims: a Prospective, Exploratory and Interventional Clinical Trial
Brief Title: Re-Step: Dynamic Balance Treatment of Gait for Acquired Brain Injury (ABI) Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-9
Record Dates: First submitted 2014-07-24; First posted 2014-08-13 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Acquired Brain Injury
Keywords: Postural balance; Motor Learning and Motor Control; Community integration; Quality of life; Functional ambulation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Re-Step (Experimental): The system consists of a pair of special shoes which sole height and angles change in a specific given order, thereby facilitating motor learning and problem solving in real time.
  This unpredictable change will introduce a situation of necessary adaptation to keep balance.
  Interventions: Device: Re-Step

INTERVENTIONS:
Device: Re-Step — Research Group:
  Each session begins with a warm-up exercise, muscle stretching, and strengthening exercises: duration 10 minutes.
  Afterwards, walking exercises for 40 minutes with Re-Step according to a program individually tailored and progressing with the training. Progress is shown by an increased range of tilting of the shoe and speed of changes, according to the individual ability of each patient.
  At the end of the session 10 min of cool-down exercises
  22 training sessions of 60 minutes each, twice a week.
  Other Names: Step of Mind's Re-Step System shoes

SUMMARY:
The purpose of this study is to:

1. Test the walking functionality of people following Acquired brain injury (ABI)
2. Suggesting a new treatment for their walking impairments
3. Follow-up of motor learning ability and balance after intervention within this population

The investigators intend to target dynamic stability and gait after ABI, in a group of individuals with ABI who have persistent balance and mobility deficits despite being able to walk independently and having high scores on standard clinical balance measures.

Interventions: Training with Re-Step system shoes.

In this study there is no control group.

DETAILED DESCRIPTION:
Study design:

Type of research: Prospective, exploratory, clinical, interventional trial

Specific objectives are:

To explore the efficacy of Re-step rehabilitation technology to improve dynamic balance in the gait of people after Acquired Brain Injury (ABI).

The investigators suggest a new technology of intervention that will induce unexpected changes of underfoot slopes, with Re-Step shoes, during walking and will force the central nervous system (CNS) to react and solve walking problems in real-time.

The investigators propose that the new approach will have a significant motor function improvement on balance in gait, transferred to real environmental settings and be retained for long periods of time.

Research methods:

Subjects:

A total of 40 subjects of ABI victims will be studied in one treatment group-Re-Step shoes walking training

Time flow protocol:

Participants will be approached using a database of hospitalized patients of Reuth Rehabilitation Hospital (Tel-Aviv, Israel) and through a call for participation placed in a newspaper.

Subjects will be recruited according to inclusion/exclusion criteria, after medical examination and given consent of participation.

Tests and measures (see outcome measures) will be applied to measure changes:

* T1 - before starting the intervention to form a baseline
* T2 - after 20 sessions of intensive treatments 60 min each, 2 sessions a week.
* T3 - 6 months after T2, a period of normal daily schedule of subjects, with no interventions, to examine for retainment of training results.

The treatments will start in a week from T1; the T2 will be performed in a week after training was completed; T3 will be performed 6 months (take or leave 2 weeks) after T2.

ELIGIBILITY:
Inclusion Criteria:

* At least one year after the Acquired brain injury.
* Age 18 to 80 years
* Independent walking ability for at least 10 meters
* Patients who permanently use medications that have not been changed during the past month and with no further changes expected during the research
* At least 19 points on the MoCA test

Exclusion Criteria:

* Presence of degenerative neurological disability that is not secondary to the acquired brain injury
* Other disabilities such as - severe back pain, radical active lumbosacral radicular pain, leg muscle pain, peripheral neuropathy, post-polio syndrome, rheumatic illnesses, previous orthopedic disabilities preceding or at the time of the injury that could affect the ability and pattern of walking, depression, and other neurotic syndromes including post-traumatic depression and post-traumatic stress disorder (PTSD) at a medium level or higher, chronic alcoholism and use of drugs.
* Unstable state of health such as heart disease, respiratory insufficiency, peripheral vascular disease, acquired brain injury that has impaired walking ability
* Inability to persevere and cooperate in the series of tests and the follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Community Balance & Mobility Scale (CB&M); Change from base line after intervention is being assessed | Measuring mobility ability and balance at base line and changes after intervention; and changes and rtainment of achievments 6 months of no intervention
  CB&M was designed to evaluate balance and mobility in patients who, although ambulatory, have balance impairments that reduce their full engagement in community living. 13 items of dynamic balance are graded 0-5 by a physiotherapist. The CB&M is a reliable and valid clinical outcome measure for evaluating change in ability in the higher functioning ambulatory patients with TBI.

SECONDARY OUTCOMES:
10 Meter walk Test (10MWT) | Measuring at base line; change immediately after intervention, and changes and retainments of achievments after 6 months
  Assesses walking speed in meters per second over a short duration. The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed). The distance covered is divided by the time it took the individual to walk that distance.
Montreal Cognitive Assessment (MoCA) | Recruitment stage
  Widely used method for assessing cognitive mental status both in clinical practice and in research.
  It is a brief, standardized method to grade patients' cognitive mental status. It assesses orientation, attention, immediate and short-term recall, language, and the ability to follow simple verbal and written commands. It provides a total score that places the individual on a scale of cognitive function.
  The MoCA test has a high sensitivity for detecting cognitive dysfunction.
fMRI functional magnetic Resonance Imaging; Change from base line after intervention is being assessed | Base line brain activity; change after treatment; and change after 6 months with no interventions
  Functional magnetic resonance imaging or functional MRI (fMRI) is a functional neuroimaging procedure using MRI technology that measures brain activity by detecting associated changes in blood flow. This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bar-Haim, PhD; PT, Principal Investigator — The Laboratory for Rehabilitation and Motor Control of Walking Faculty of Health Sciences at Ben-Gurion University of the Negev Israel; Jean-Jacques Vatine, Dr., Study Director — Reuth Rehabilitation Hospital Tel-Aviv Israel.
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

REFERENCES:
- [Derived] Joubran K, Bar-Haim S, Shmuelof L. Dynamic balance recovery in chronic acquired brain injury participants following a perturbation training. Int J Rehabil Res. 2021 Dec 1;44(4):350-357. doi: 10.1097/MRR.0000000000000485. PMID 34739006